CLINICAL TRIAL: NCT02379819
Title: Nucleus Hybrid L24 Implant System: New Enrollment Study
Brief Title: Hybrid L24 New Enrollment Post Approval Study
Acronym: HNE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cochlear (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAM-5573-HYB-PMA
Record Dates: First submitted 2015-01-29; First posted 2015-03-05 (Estimated); Results first posted 2023-03-13 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-02

CONDITIONS: High Frequency Sensorineural Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes

ARMS (1):
- Nucleus Hybrid L24 Implant (Experimental): Adults age 18 and over who meet FDA criteria for unilateral implantation with the Nucleus Hybrid L24 Implant.
  Interventions: Device: Nucleus Hybrid L24 Implant

INTERVENTIONS:
Device: Nucleus Hybrid L24 Implant

SUMMARY:
This study evaluates the long term safety and effectiveness of the Nucleus Hybrid L24 Implant in a group of newly implanted adults.

ELIGIBILITY:
Inclusion Criteria:

Ear to Be Implanted:

* Normal to moderate hearing loss in the low frequencies with severe to profound mid to high frequency hearing loss in the ear to be implanted
* CNC word recognition of 10-60% in the ear to be implanted

Contralateral Ear:

* Moderately severe to profound mid to high frequency hearing loss in the contralateral ear
* CNC word recognition equal to or better than that in the ear to be implanted but not more than 80% correct

Exclusion Criteria:

* not proficient in English
* unwilling and/or unable to comply with the test protocol
* deafness due to lesions of the acoustic nerve or central auditory pathway.
* active middle-ear disease, with or without tympanic membrane perforation.
* absence of cochlear development.
* duration of severe to profound hearing loss of 30 years or greater

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2022-04-14 (Actual); Study Completion 2022-04-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Kaplan, MD, Principal Investigator — Greater Baltimore Medical Center
Locations (19):
- United States (19):
  - Arizona Ear Center, Phoenix, Arizona
  - Kaiser Permanente South Sacramento, Sacramento, California
  - University of Colorado Hospitals, Aurora, Colorado
  - Denver Ear Associates, Englewood, Colorado
  - Rocky Mountain Ear Center, Englewood, Colorado
  - University of Miami, Miami, Florida
  - NorthShore University Health System, Northbrook, Illinois
  - University of Iowa, Iowa City, Iowa
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Michigan Ear Institute, Farmington Hills, Michigan
  - Midwest Ear Institute, Kansas City, Missouri
  - The University of Cincinnati, Cincinnati, Ohio
  - Ohio Ear Institute, Westerville, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Pittsburgh Ear Associates, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Ear Institute of Texas, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No
Cochlear do not have an approved platform for public sharing of IPD collected in this study. Data may be provided to individual researchers on request.

REFERENCES:
- [Derived] Reinhart PN, Parkinson AJ, Dunn CC, Gantz BJ. Factors Affecting Audiometric and Speech Perception Outcomes in Hybrid Cochlear Implant Recipients. Laryngoscope. 2025 Oct 8. doi: 10.1002/lary.70195. Online ahead of print. PMID 41059917
- [Derived] Reinhart P, Parkinson A, Gifford RH. Hybrid Cochlear Implant Outcomes and Improving Outcomes With Electric-Acoustic Stimulation. Otol Neurotol. 2024 Dec 1;45(10):e749-e755. doi: 10.1097/MAO.0000000000004305. PMID 39514431

RESULTS

PARTICIPANT FLOW:
Groups:
- Nucleus Hybrid L24 Implant: Adults age 18 and over who meet FDA criteria for unilateral implantation with the Nucleus Hybrid L24 Implant.
  Nucleus Hybrid L24 Implant
Period: Overall Study
Arm/Group | Nucleus Hybrid L24 Implant
Started | 52
Completed | 38
Not Completed | 14
Not completed — Withdrawal by Subject | 10
Not completed — Death | 2
Not completed — Lack of Efficacy | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Nucleus Hybrid L24 Implant
Number analyzed (Participants) | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.9 (15.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 25
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 52

OUTCOME MEASURES:

1. Primary Outcome: Change in Consonant-Nucleus-Consonant (CNC) Word Recognition in Quiet for the Two Listening Conditions: Implant Ear Alone and When Using Both Ears Together From Pre-operatively Through 3 Years Post-activation of the Device
Description: The CNC Words test consists of 10 recorded lists of 50 monosyllabic words in CD format. For this study, two lists will be administered in quiet at a level equal to 60 dBA in the sound field and recorded as a total number of words correct, which will be expressed as a percentage correct for this study. The CNC word test has a score range of 0-100% with higher values indicating better scores.
Time Frame: From pre-operatively through 3 years post-activation of the device
Population: Data was not collected for all 52 participants at all of the time points. At 2 years post-activation, one participant doesn't have a bilateral speech score.
Measure: Mean (95% Confidence Interval); unit: percentage of correct words
Arm/Group | Nucleus Hybrid L24 Implant
Number analyzed (Participants) | 50
percentage of correct words
  Unilateral condition at 3 months post-activation | 31.3 [25.4 to 37.3]
  Unilateral condition at 6 months post-activation: number analyzed (Participants) | 49
  Unilateral condition at 6 months post-activation | 35.2 [29.3 to 41.1]
  Unilateral condition at 1 year post-activation: number analyzed (Participants) | 48
  Unilateral condition at 1 year post-activation | 35.8 [29.6 to 41.9]
  Unilateral condition at 2 years post-activation: number analyzed (Participants) | 47
  Unilateral condition at 2 years post-activation | 35.3 [29.2 to 41.5]
  Unilateral condition at 3 years post-activation: number analyzed (Participants) | 38
  Unilateral condition at 3 years post-activation | 36.8 [29.7 to 44.0]
  Bilateral condition at 3 months post-activation | 26.8 [22.2 to 31.5]
  Bilateral condition at 6 months post-activation: number analyzed (Participants) | 49
  Bilateral condition at 6 months post-activation | 29.7 [24.6 to 34.8]
  Bilateral condition at 1 year post-activation: number analyzed (Participants) | 48
  Bilateral condition at 1 year post-activation | 31.1 [26.4 to 35.9]
  Bilateral condition at 2 years post-activation: number analyzed (Participants) | 46
  Bilateral condition at 2 years post-activation | 32.4 [26.8 to 38.0]
  Bilateral condition at 3 years post-activation: number analyzed (Participants) | 38
  Bilateral condition at 3 years post-activation | 32.5 [26.7 to 38.3]

2. Primary Outcome: Number of Device or Procedure Related Adverse Events
Time Frame: Up to 5 years post-activation of the device
Population: Related AEs were reported up to 3 years with some participants up to 5 years as the protocol was amended from 5 to 3 year follow-up in 2022.
  The data include all related AEs reported.
Measure: Number; unit: Number of events
Arm/Group | Nucleus Hybrid L24 Implant
Number analyzed (Participants) | 52
Number of events
  Total number of device or procedure related adverse event | 98
  Number of serious device or procedure related adverse event | 1

3. Secondary Outcome: Change in AzBio Sentence Recognition in Noise in the Best Unilateral Condition
Description: The AzBio Sentence Tests consists of 15 lists of 20 sentences each. AzBio sentences are spoken by different talkers in a conversational style with limited contextual cues that the listener can use to predict or 'fill in' unintelligible words. Each list includes 5 sentences from 4 different male and female speakers. Each word in the sentence counts toward the overall score and the resulting score is presented in percent correct. The AzBio sentence test has a score range of 0-100% with higher values indicating better scores.
Time Frame: Pre-operatively, up to 3 years post-activation of the device
Population: Data was not collected for all 52 participants at all of the time points. At 1 year post-activation, one participant completed the testing at +10 dB SNR (decibel signal to noise ratio) instead of +5 dB SNR which is what is reported on.
Measure: Mean (95% Confidence Interval); unit: percentage of correct words
Arm/Group | Nucleus Hybrid L24 Implant
Number analyzed (Participants) | 50
percentage of correct words
  At 3 months post-activation | 18 [11.5 to 24.6]
  At 6 months post-activation: number analyzed (Participants) | 49
  At 6 months post-activation | 24.4 [17.4 to 31.3]
  At 1 year post-activation: number analyzed (Participants) | 47
  At 1 year post-activation | 21.5 [15.2 to 27.9]
  At 2 years post-activation: number analyzed (Participants) | 47
  At 2 years post-activation | 23.7 [17.4 to 29.9]
  At 3 years post-activation: number analyzed (Participants) | 38
  At 3 years post-activation | 17.8 [9.1 to 26.5]

ADVERSE EVENTS:
Time Frame: Up to 5 years
Description: Device and procedure related adverse events are reported. The related AEs were reported up to 3 years with some patients up to 5 years as the protocol was amended from 5 to 3 year follow-up in 2022. Two participants passed away but the cause of death was not related to the device or procedure.
Arm/Group | Nucleus Hybrid L24 Implant
All-Cause Mortality (participants affected / at risk) | 2/52
Serious Adverse Events (participants affected / at risk) | 1/52
Other Adverse Events (participants affected / at risk) | 35/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nucleus Hybrid L24 Implant (N=52)
Explantation at patient's request due to sound quality (Ear and labyrinth disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nucleus Hybrid L24 Implant (N=52)
Profound hearing loss (Ear and labyrinth disorders) | 20 (20)
New or worsened tinnitus (Ear and labyrinth disorders) | 8 (8)
Vertigo/dizziness (Ear and labyrinth disorders) | 18 (20)
Skin irritation due to externals (General disorders) | 5 (5)
Pain in implanted ear (Ear and labyrinth disorders) | 4 (5)
Nausea/vomiting (Gastrointestinal disorders) | 4 (4)
Sound quality issue (Product Issues) | 3 (3)
Taste/Tongue disturbance (General disorders) | 3 (4)
Ear numbness (General disorders) | 3 (3)
Small parts hazard (Product Issues) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The aggregate data resulting from this study will be the proprietary information of the Sponsor and may be made public after all data have been analyzed and the study results are available. None of the data resulting from this study will be allowed to be presented or published in any form, by the Investigator or any other person, without the prior written approval of the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2022-04-30): https://cdn.clinicaltrials.gov/large-docs/19/NCT02379819/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-30): https://cdn.clinicaltrials.gov/large-docs/19/NCT02379819/SAP_001.pdf